CLINICAL TRIAL: NCT05077137
Title: A Feasibility Study Utilizing Immune Recall to Increase Response to Checkpoint Therapy
Acronym: TdVax
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108367
Record Dates: First submitted 2021-09-13; First posted 2021-10-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Td Vaccine (Experimental): The first 15 subjects enrolled will receive the Td (tetanus diphtheria) vaccine at cycle 4 of IO therapy. The Td vaccine is administered as 0.5 mL intramuscular injection in the extremity (thigh or upper arm) in closest proximity to the largest tumor.
  Interventions: Biological: Tetanus Diptheria Vaccine
- IPOL Vaccine (Experimental): Subjects 16 through 25 will receive the IPOL (polio booster) vaccine at cycle 4 of IO therapy. The IPOL vaccine is administered as 0.5 mL intramuscular or subcutaneous injection in the extremity (thigh or upper arm) in closest proximity to the largest tumor
  Interventions: Biological: Polio Boost Immunization

INTERVENTIONS:
Biological: Tetanus Diptheria Vaccine — tetanus and diphtheria toxoids
  Other Names: Tenivac
  Arms: Td Vaccine
Biological: Polio Boost Immunization — trivalent inactivated polio vaccine
  Other Names: IPOL
  Arms: IPOL Vaccine

SUMMARY:
The purpose of this study is to determine the safety and feasibility of administering the Tetanus Diptheria Vaccine (Td) or Polio Boost Immunization (IPOL) to patients with metastatic melanoma who are receiving immune checkpoint inhibitor (IO) therapy per standard of care. Subjects will have the vaccine at cycle 4 of IO therapy and will have research blood and tissue samples collected prior to starting IO therapy, at cycle 4 prior to vaccine administration, and at 12-17 days post vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced metastatic melanoma
2. Male or female participants who are at least 18 years of age on the day of signing informed consent
3. Participants must be planned or scheduled by their treating physician to receive PD-1 therapy or PD-1 plus anti CTLA-4 therapy as standard of care
4. Participant (or legally acceptable representative if applicable) provides written informed consent for the trial
5. Participant must have at least 1 lesion that is at least 8 mm in size and is cutaneous, subcutaneous, palpable, or amenable to ultrasound guided core biopsy. The lesion chosen for biopsy can also be a target lesion but does not have to be a target lesion
6. Adequate organ function as defined below. Standard of care labs drawn within 45 days prior to consent may be used for the purposes of determining eligibility

   1. ANC >/= 1500/uL
   2. platelets >/=100,000/uL
   3. Hemoglobin >/= 9.0 g/dL

Exclusion Criteria:

1. Uveal or mucosal melanoma
2. Any women known to be pregnant or breastfeeding
3. Any prior systemic therapy for metastatic melanoma (prior surgery is allowed)
4. Known diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone or equivalent), or any other form of immunosuppressive therapy within 7 days prior to first research biopsy
5. Patients with symptomatic CNS metastases and/or carcinomatous meningitis

   a) Patients with asymptomatic, stable CNS metastases are allowed provided that they are not on >10mg prednisone daily
6. History of or active (non-infectious) pneumonitis that required steroids
7. Active infection requiring systemic therapy
8. Known history of Human Immunodeficiency Virus (HIV) infection
9. Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. NOTE: no testing for Hepatitis B or Hepatitis C is required
10. Known history of active TB (Bacillus Tuberculosis)
11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with subject's participation for the full duration of the study, or make it not in the best interest of the subject to participate, in the opinion of the treating physician
12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
13. History of allogenic tissue or solid organ transplant
14. History of allergic reaction to IPOL or Td vaccine
15. Receipt of Td vaccine within 30 days prior to starting IO therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects out of the proposed 25 that successfully receive the vaccine after 4 cycles of IO therapy | informed consent through date of vaccine (est apx 4-5 months)
  Evaluable patients are defined as those who receive four cycles of IO therapy and then receive a Td or IPOL vaccine
Safety, as measured by the change in the number and severity of adverse events deemed related to the vaccine or study procedures (blood draw and biopsies) | Baseline, cycle 4 of IO therapy (apx 12-16 weeks), 12-17 days post vaccine, SOC scan following vaccine (apx 8-12 weeks post vaccine)
  Adverse events will only include those that are determined to be related to the study vaccine or study procedures (blood draw and biopsies)

SECONDARY OUTCOMES:
Preliminary efficacy, as measured by objective response rate | up to 36 months
  Number of patients that experience tumor response vs. stable disease vs. progression as determined by PI assessment of standard of care scans

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Beasley, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be used internally by the study team